CLINICAL TRIAL: NCT02996786
Title: Effects of Danggui Buxue Tang on Blood Biochemical Parameters in Male Recreational Runners
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MOST 106-2410-H-037-007-MY3
Record Dates: First submitted 2016-12-11; First posted 2016-12-19 (Estimated); Last update posted 2018-04-20 (Actual); Status verified 2016-11

CONDITIONS: Sports Anemia; Inflammation; Oxidative Stress; Iron Deficiency; Hemolysis; Fatigue
MeSH Terms: conditions — Inflammation; Iron Deficiencies; Hemolysis; Fatigue | interventions — danggui buxue decoction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Danggui Buxue Tang group (Experimental): Danggui Buxue Tang group receive orally supplementation of 7.5 g/day of Danggui Buxue Tang for 10 days
  Interventions: Dietary Supplement: Danggui Buxue Tang
- Placebo group (Placebo Comparator): Placebo group receive orally supplementation of 7.5 g/day of placebo for 10 days
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Danggui Buxue Tang — Danggui Buxue Tang purchased from Kaiser Pharmaceutical
  Arms: Danggui Buxue Tang group
Other: Placebo — Consisting of corn starch and carboxymethyl cellulose
  Arms: Placebo group

SUMMARY:
The aim of this study is to examine the beneficial effects of Danggui Buxue Tang on blood biochemical parameters in male recreational runners.

DETAILED DESCRIPTION:
1. Male recreational runners would be recruited by community websites or email. After completely introducing the study, the participants would be requested to sign informed consent.
2. The participants would perform maximal oxygen consumption test prior to the supplementation. The participants would be supplemented with either Danggui Buxue Tang or placebo for a week before performing the 13-km run. A total of 4 times blood collection (before supplementation, immediate after running, 1 day and 3 days after running) would be performed for evaluating the effect of Danggui Buxue Tang on blood biochemical parameters.

ELIGIBILITY:
Inclusion Criteria:

* The participants should have the experience finishing 10-km run but without the experience of attending a marathon run.

Exclusion Criteria:

* Participants suffering from anemia (Hb <13 g/dL), taking usual supplements, medication, alcohol or not feeling comfortable.

Ages: 20 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Hematological parameters | Through study completion, an average of 1 year
  Complete blood counts and serum haptoglobin and erythropoietin
Iron status | Through study completion, an average of 1 year
  Serum iron, ferritin, transferrin and hepcidin
Oxidative stress | Through study completion, an average of 1 year
  Thiobarbituric acid reactive substances, superoxide dismutase, catalase, and glutathione peroxidase
Inflammatory response | Through study completion, an average of 1 year
  High-sensitivity c-reactive protein, Tumor necrosis factor-alpha, and interleukin-6

SECONDARY OUTCOMES:
Running time | Through study completion, an average of 1 year
  The completion time for a 13-km run

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Medical University, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No